CLINICAL TRIAL: NCT06529185
Title: Effect of Breather on Ventilatory and Vascular Function in Chronic Obstructive Pulmonary Disease Patients with Intermittent Claudication.
Brief Title: Effect of Breather in COPD Patients with Intermittent Claudication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Medhat Mohamed Ali Farahat, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Breather on COPD with IC
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-10

CONDITIONS: COPD; PAD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Drug Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): This group include 30 patients with COPD and intermittent claudication. These patients can receive aerobic exercise (by applying treadmill exercise for 20 min) and inspiratory muscle training (by using The BREATHER device with Light/Medium resistance for 3-5 sets /session), for 4 weeks (3 sessions per week) and pursed lip breathing.
  Interventions: Device: The BREATHER
- control group (Active Comparator): This group include 30 patients with COPD and intermittent claudication. These patients can receive pursed lip breathing and aerobic exercise (by applying treadmill exercise for 20 min) with the usually pharmacological treatment, for 4 weeks (3 sessions per week).
  Interventions: Drug: pharmacological treatment

INTERVENTIONS:
Device: The BREATHER — The BREATHER is Light/Medium resistance inspiratory muscle trainer which has significance role in increasing inspiratory muscle strength and endurance which could result in a decreased sensation of dyspnea
  Other Names: experimental group
  Arms: treatment group
Drug: pharmacological treatment — patient will receive the usually pharmacological treatment.
  Other Names: control group
  Arms: control group

SUMMARY:
The aim of this study To show the effect of breather on ventilatory and vascular function in COPD patient with intermittent claudication.

DETAILED DESCRIPTION:
recent researches show that COPD patients have risk of developing peripheral arterial disease (PAD) which represented on patient by intermittent claudication inspiratory muscle trainer as the breather device show increasing in inspiratory muscle strength and endurance; reduction of dyspnea; and improving of exercise tolerance .

Because of all this things this study tends to show the effect of the breather on ventilatory and vascular function in COPD patient with intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

* sixty male patients with diagnosed with grade I and grade II COPD their ages ranged between 55-60years
* All patients will be clinically and medically stable when attending the study.
* Body mass index (BMI) is 18.5 to 24.9 kg/m2.
* History of unilateral exertional leg pain,
* Ambulation during a graded treadmill test limited by leg pain consistent with intermittent claudication (stage II of the fontaine classification of pad),
* And an ankle-brachial index (ABI) of 0.90 or lower at rest or 0.73 or lower after exercise.

Exclusion Criteria:

* cardiovascular insufficiency,
* Recent myocardial infarction,
* heart failure,
* arrhythmia,
* DVT,
* Intracranial hypertension,
* Pneumonia,
* kidney failure,
* fractures,
* uncooperative patients,
* cognitive impairment preventing a patient from participation in exercises.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Ventilatory function: by spirometry test | 4 weeks
  Spirometry is a physiological test that measures the ability to inhale and exhale air relative to time.
Vascular function: by doppler ultrasound | 4 weeks
  Doppler ultrasound is a simple and non-invasive and method for the evaluation of early atherosclerosis. It can be used as a screening program for PAD in populations with high risk for atherosclerosis.

SECONDARY OUTCOMES:
Functional capacity assessment: by 5 repetitions sit to stand test (5R-STS) | 4 weeks
  (5R-STS) test is an objective test of functional impairment commonly used in various diseases including COPD which is used to measure the severity of disease and to monitor recovery.
Treadmill exercise testing | 4 weeks
  The results of the tests will be expressed in units of distance that will be walked up to the claudication pain (initial claudication distance) and the maximally tolerated claudication pain (maximal claudication distance).

CONTACTS AND LOCATIONS:
Overall Officials: Zahra M Serry, Assist.Prof, Study Director — Cairo University; MARWA M ELSAYED, Assist.Prof, Study Director — Cairo University; Amira I Almeldin, Assist.Prof, Study Director — Cairo University; reem M farahat, student, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaumont M, Forget P, Couturaud F, Reychler G. Effects of inspiratory muscle training in COPD patients: A systematic review and meta-analysis. Clin Respir J. 2018 Jul;12(7):2178-2188. doi: 10.1111/crj.12905. Epub 2018 May 23. PMID 29665262
- [Background] Pinto B, Correia MV, Paredes H, Silva I. Detection of Intermittent Claudication from Smartphone Inertial Data in Community Walks Using Machine Learning Classifiers. Sensors (Basel). 2023 Feb 1;23(3):1581. doi: 10.3390/s23031581. PMID 36772621
- [Background] Terzikhan N, Lahousse L, Verhamme KMC, Franco OH, Ikram AM, Stricker BH, Brusselle GG. COPD is associated with an increased risk of peripheral artery disease and mortality. ERJ Open Res. 2018 Dec 21;4(4):00086-2018. doi: 10.1183/23120541.00086-2018. eCollection 2018 Oct. PMID 30588480
- [Derived] Elsayed MM, Farahat RM, Serry ZH, Almeldin AI. Inspiratory Muscle Training and Aerobic Exercise Affect Chronic Obstructive Pulmonary Disease Patients With Intermittent Claudication: A Randomized Controlled Trial. Physiother Res Int. 2026 Jan;31(1):e70130. doi: 10.1002/pri.70130. PMID 41287032